CLINICAL TRIAL: NCT00460187
Title: Evaluating the Use of the FiberNet Embolic Protection System in Carotid Artery Stenting: The EPIC US Pivotal Study.
Brief Title: EPIC US Pivotal Study
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumen Biomedical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90-1145
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Percutaneous Intervention of the Carotid Arteries.
Keywords: carotid artery, distal protection device, carotid stenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Percutaneous intervention of the carotid artery

SUMMARY:
Multicenter, prospective, pivotal study designed to demonstrate the safety and efficacy of the Lumen Biomedical, Inc. FiberNet® Embolic Protection System as an adjunctive device during carotid artery percutaneous intervention in high surgical risk patients.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the high surgical risk criteria.
* Symptomatic with atherosclerotic stenosis ≥ 50% or asymptomatic with atherosclerotic stenosis ≥ 70% of the carotid artery by NASCET Criteria.

Exclusion Criteria:

* Prior stenting of ipsilateral carotid.
* Planned treatment of contralateral carotid within 30 days.
* Experienced a myocardial infarction within the last 14 days.
* Undergone an angioplasty or PTCA/PTA procedure within the past 48 hours.
* Undergone cardiac surgery within the past 60 days.
* Suffered a stroke within the past 14 days.
* Suffered a transient ischemic neurological attack (TIA) or amaurosis fugax within the past 48 hours.
* Abnormal baseline blood counts; platelets <50,000 or >700,000/mm3 or WBC count < 3 x103/uL.
* Intracranial stenosis that exceeded the severity of an extracranial stenosis.
* Total occlusion of the target vessel.
* Lesion within 2cm of the ostium of the common carotid artery.
* A stenosis that is known to be unsuitable for stenting
* Serial lesions that requires more than one stent to cover entire lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2007-03; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The rate of all death, all stroke and myocardial infarction within 30 days of the procedure.

SECONDARY OUTCOMES:
Secondary Endpoints are: all death and all stroke rates, non-stroke neurological event rates, technical success rates, procedural success rates, and access site complication rates.

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Bacharach, MD, Principal Investigator — Heart Hospital of South Dakota; Subbarao Mylavarapu, MD, Principal Investigator — Hoag Hospital
Locations (2):
- United States (2):
  - Hoag Hospital, Newport Beach, California
  - Heart Hospital of South Dakota, Sioux Falls, South Dakota

REFERENCES:
- See also: Lumen Biomedical website — http://www.lumenbio.com